CLINICAL TRIAL: NCT06916741
Title: Examining the Effect of a Sacral Lift on Femoral Vein Size and Exposure in the Emergency Department
Brief Title: Effect of a Sacral Lift on Femoral Vein Size and Exposure
Acronym: Sacral Lift
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Dr. Dhimitri Nikolla, EM Core Faculty / Research Director, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: Sacral Lift
Record Dates: First submitted 2025-02-20; First posted 2025-04-08 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Femoral Artery; Cannulation
Keywords: femoral artery; ultrasound; femoral vein; sacral lift; cannulation
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: The study design is a single-blinded, randomized (nested randomization of leg position and sacral lift sequence within randomized leg sequence [i.e., left, right]) cross-over study.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacral Lift First (Experimental): Femoral vein measurements are first collected using a sacral lift, then collected again without using a sacral lift.
  Interventions: Diagnostic Test: Ultrasound with Sacral lift
- Sacral Lift Second (Experimental): Femoral vein measurements are first collected without using a sacral lift, then collected again using a sacral lift.
  Interventions: Diagnostic Test: Ultrasound with Sacral lift

INTERVENTIONS:
Diagnostic Test: Ultrasound with Sacral lift — Intervention includes using a sacral lift during ultrasound to collect femoral vein measurements.

SUMMARY:
The goal of this clinical trial is to learn if a sacral lift can improve femoral vein size and exposure, which may be clinically helpful during femoral vein cannulation among emergency department patients. The main questions it aims to answer are:

Does a sacral lift increase femoral vein size compared to no sacral lift in both straight and frog-leg positions? Does a sacral lift improve femoral vein exposure (reduce overlap by the femoral artery) compared to no sacral lift in both straight and frog-leg positions? Researchers will compare femoral vein size and exposure measurements with and without a sacral lift in both straight and frog-leg leg positions to see if the sacral lift improves vein size and reduces artery overlap.

Participants will:

Undergo femoral vein ultrasound scans. Maintain a straight leg position with and without a sacral lift. Maintain a frog-leg position with and without a sacral lift.

DETAILED DESCRIPTION:
This study is a clinical trial designed to investigate the effectiveness of a sacral lift in improving femoral vein size and exposure. If a sacral lift improves femoral vein size and/or exposure, it may improve the success rate of femoral vein cannulation, a critical resuscitative procedure. Femoral vein cannulation can be difficult when the vein is overlapped by the femoral artery. While positioning the leg in abduction with external rotation and knee flexion ("frog-leg" position) is known to improve femoral vein exposure, this study explores the potential added benefit of a sacral lift (a gel pad placed under the sacrum). The study will focus on emergency department patients who frequently require this procedure.

The primary purpose is to determine if the addition of a sacral lift improves femoral vein size and exposure, thereby potentially facilitating easier and more successful cannulation. The study will address the following key questions:

Does the use of a sacral lift significantly increase femoral vein diameter compared to no sacral lift, in both straight leg and frog-leg positions?

Does the use of a sacral lift significantly improve the visualization of the femoral vein (reduce femoral artery overlap) compared to no sacral lift, in both straight leg and frog-leg positions?

The study will employ a comparative design, measuring femoral vein size and assessing the degree of femoral artery overlap with and without a sacral lift, in both straight leg and frog-leg positions. This will allow researchers to directly compare the impact of the sacral lift on these critical factors affecting cannulation success. The findings will provide valuable data for optimizing the technique of femoral vein cannulation and improving outcomes in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult emergency department patients.

Exclusion Criteria:

* <18 or >85 years-old
* Anyone with a history of: deep venous thrombosis (DVT), May-Thurner syndrome, lower extremity vein harvesting, arterial or venous surgery of the lower leg (e.g., peripheral arterial stent placement or sclerotherapy of lower extremity varicose veins), or peripheral vascular disease.
* Anyone with a medical condition that could impact their physical ability to lay supine or abduct and externally rotate their hips safely (e.g., hip fracture).
* Anyone whose femoral vessels cannot be clearly identified using a linear transducer
* Anyone whose femoral vein is not compressible on the study ultrasound (indicating a DVT). If 100% of the femoral vein is already exposed from under the femoral artery with a straight leg (right or left), the patient will be excluded from the study.
* Vulnerable populations such as pregnant women and those who cannot consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Potential effect of a sacral lift on femoral vein cross-sectional area | From enrollment to end of ultrasound measurements, expected to take up to one hour
  Our objective is to use ultrasound measurements to compare femoral vein cross-sectional area in centimeters squared (cm^2) within each subject with and without a sacral lift.

SECONDARY OUTCOMES:
Potential effect of a sacral lift on measurements of femoral vein diameter | From enrollment to end of ultrasound measurements, expected to take up to one hour
  Our objective is to use ultrasound measurements to compare femoral vein diameter (from the medial to lateral wall of the femoral vein) in centimeters between within each subject with and without a sacral lift.
Potential effect of a sacral lift on measurements of femoral vein exposure | From enrollment to end of ultrasound measurements, expected to take up to one hour
  Our objective is to use ultrasound measurements to compare femoral vein exposure (proportion of the width of the femoral vein not overlapped by the femoral artery: width of femoral vein in centimeters - width of femoral vein overlapped by femoral artery in centimeters / width of femoral vein in centimeters *100) between within each subject with and without a sacral lift.
Potential effect of a sacral lift on measurements of femoral vein depth | From enrollment to end of ultrasound measurements, expected to take up to one hour
  Our objective is to use ultrasound measurements to compare femoral vein depth (from skin to most superficial wall) in centimeters between within each subject with and without a sacral lift.

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator Dhimitri Nikolla, DO, MS, FACEP, FACOEP, Principal Investigator — Allegheny Health Network
Locations (1):
- Saint Vincent Hospital, Erie, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
It is not necessary for the scope of the study to share IPD.

REFERENCES:
- [Background] Stone MB, Price DD, Anderson BS. Ultrasonographic investigation of the effect of reverse Trendelenburg on the cross-sectional area of the femoral vein. J Emerg Med. 2006 Feb;30(2):211-3. doi: 10.1016/j.jemermed.2005.05.022. PMID 16567260
- [Background] Kim W, Chung RK, Lee GY, Han JI. The effects of hip abduction with external rotation and reverse Trendelenburg position on the size of the femoral vein; ultrasonographic investigation. Korean J Anesthesiol. 2011 Sep;61(3):205-9. doi: 10.4097/kjae.2011.61.3.205. Epub 2011 Sep 23. PMID 22025941
- [Background] Kim JT, Lee NJ, Na HS, Jeon Y, Kim HS, Kim CS, Kim SD. Ultrasonographic investigation of the effect of inguinal compression on the cross-sectional area of the femoral vein. Acad Emerg Med. 2008 Jan;15(1):101-3. doi: 10.1111/j.1553-2712.2007.00018.x. PMID 18211323
- [Background] Suk EH, Kim DH, Kil HK, Kweon TD. Effects of reverse Trendelenburg position and inguinal compression on femoral vein cross-sectional area in infants and young children. Anaesthesia. 2009 Apr;64(4):399-402. doi: 10.1111/j.1365-2044.2008.05815.x. PMID 19317705
- [Background] Kim JT, Park CS, Kim HJ, Lee JM, Kim HS, Kim CS, Kim SD. The effect of inguinal compression, Valsalva maneuver, and reverse Trendelenburg position on the cross-sectional area of the femoral vein in children. Anesth Analg. 2009 May;108(5):1493-6. doi: 10.1213/ane.0b013e31819bccc7. PMID 19372327
- [Background] Werner SL, Jones RA, Emerman CL. Effect of hip abduction and external rotation on femoral vein exposure for possible cannulation. J Emerg Med. 2008 Jul;35(1):73-5. doi: 10.1016/j.jemermed.2007.03.023. Epub 2007 Aug 29. PMID 17976787
- [Background] Ahn JH, Park J, Song IS, Kim KA, Park J, Min JJ, Kim CS, Lee JH. The angle range of leg abduction with external hip rotation which can minimize femoral artery and vein overlap in pediatric patients. Paediatr Anaesth. 2019 Apr;29(4):361-367. doi: 10.1111/pan.13603. Epub 2019 Mar 21. PMID 30735284
- [Background] Read H, Holdgate A, Watkins S. Simple external rotation of the leg increases the size and accessibility of the femoral vein. Emerg Med Australas. 2012 Aug;24(4):408-13. doi: 10.1111/j.1742-6723.2012.01568.x. Epub 2012 Apr 25. PMID 22862758
- [Background] Randall C, Schmeiser E, Fiers E, Little A, Dogbey G, Richardson G. Ultrasound investigation of leg position to enhance femoral vein exposure for cannulation. J Emerg Med. 2014 Aug;47(2):176-81. doi: 10.1016/j.jemermed.2014.02.001. Epub 2014 Apr 13. PMID 24725821
- [Background] Castro D, Martin Lee LM, Bhutta BS. Femoral Vein Central Venous Access(Archived). 2023 Aug 17. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK459255/ PMID 29083581